CLINICAL TRIAL: NCT03784651
Title: Metabolic and Bone Changes After Adjuvant Cancer Treatments in Early Non-metastatic Breast Cancer - a 5-year Follow-up Study.
Brief Title: Metabolic and Bone Changes After Adjuvant Cancer Treatments in Early Non-metastatic Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kristian Buch, Principal investigator, Rigshospitalet, Denmark
Other Study IDs: H-18016600
Record Dates: First submitted 2018-06-29; First posted 2018-12-24 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Bone Fracture; Glucose, High Blood; Insulin Resistance; Blood Pressure, High; Cholesterolemia
MeSH Terms: conditions — Fractures, Bone; Insulin Resistance; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer is the most common cancer type in European women. Patients treated for early non-metastatic breast cancer comprise a growing group of survivors due to early diagnosis and improved treatment. Many of these survivors experience adverse effects such as decreased bone mineral density, derangement of metabolic markers (fat, glucose, insulin) and increased blood pressure. Increasing risk of bone fracture and cardiometabolic disease (eg. diabetes mellitus type 2).

The purpose of this study is to identify mechanisms behind cardiometabolic changes that may be connected to the (neo-)adjuvant treatment. On top of this we hope to indentify potential biological markers that can help prevent development of metabolic disease.

We will be recruiting 120 post-menopausal women age 50-70 with early breast cancer and 1-2 times a year for 5 years examine bone mineral density, body composition, glucose and fat metabolism and nerve damage. A questionnaire will be used to collect information on diet, physical activity and quality of life. Derudover anvendes spørgeskemaer til at indsamle information vedrørende. This new knowledge will help clinicians start adequate preventive measures to help patients avoid cardiometabolic disease secondary to cancer treatment.

DETAILED DESCRIPTION:
Purpose and background Breast cancer is the most common cancer in Danish women, and has an average of 4,750 new cases a year (1). Patients treated for early (non-metastatic) breast cancer (EBC) comprise, due to earlier diagnosis and improved treatment, a large and growing group of cancer survivors. However, many patients experience treatment-related endocrine side-effects such as reduced bone mineral density (BMD), dyslipidemia, insulin resistance and hypertension increasing the risk of bone fractures as well risk of development of cardiometabolic disease including Type 2 diabetes (T2D).

The purpose of the study is to understand the underlying physiological and molecular mechanisms responsible for the chemotherapy-induced bone and cardiometabolic derangements to identify novel disease mechanisms as well as to identify potential biomarkers to be used for better prediction and prevention of metabolic disease.

Objectives:

In a cohort of women (n=120) with EBC to assess (WP1):

• Bone metabolism, body composition, insulin resistance, neuropathy, bone mineral density (BMD) and lung function before chemotherapy, after chemotherapy and during five years follow-up.

Background Patients treated for EBC comprise, due to earlier diagnosis and improved treatment, a large and growing group of cancer survivors. However, there might be unintended complications associated with the treatment, since patients experience treatment-related endocrine side-effects including an average weight gain of approximately 5 kg primarily reflected by an increase in fat mass and a decrease in muscle mass and thus change in body composition (2, 3). Besides less physical activity contributing to weight gain, (neo-)adjuvant chemotherapy and anti-estrogen treatment administered to prevent disease recurrence, may cause sarcopenia, increased appetite, reduced basal metabolic rate and altered whole-body metabolism (4, 5). Obesity is not only a risk factor for breast cancer development but also a risk factor for recurrence of breast cancer (6, 7). In addition to increased weight, several studies have reported increased fasting glucose, insulin and adipokine levels, increased lipids, increased insulin resistance (homeostatic model assessment (HOMA-IR)) as well as hypertension in response to chemotherapy (3, 5, 8, 9). All together these metabolic changes may induce a prediabetic phenotype associated with increased risk of developing cardiometabolic disease including Type 2 diabetes as well as cancer recurrence (10).

Patients with estrogen receptor positive early breast cancer may be sensitive to antihormonal therapy. For postmenopausal women, a common adjuvant hormonal therapy is with an aromatase inhibitor (AI) for five years (11). However, treatment with AIs is associated with reduction in BMD and increase in fracture risk due to accelerated bone resorption from estrogen suppression (12-16). Previous studies reported the highest rates of bone loss during the first year of AI treatment (17). Additionally, it has been shown that the increased bone resorption and bone loss with regard to AI can be prevented and managed with lifestyle changes, calcium and vitamin-D supplementation and the use of anti-resorptive medication (18-22).

Women with hormone receptor-positive breast cancer (BC) have an 88% 5-year survival, and if hormone-receptor-positive EBC, this is even higher and underscores the importance of ensuring that therapeutic interventions do not confer long-term morbidity.

The underlying cause for the changes in body composition during chemotherapy has not been well described and likewise has the underlying physiological and molecular mechanisms responsible for the cardio-metabolic derangements not been described either. Understanding the underlying causes and impact of treatment-related metabolic disease, will allow clinicians to initiate interventions to prevent, that these otherwise healthy women develop metabolic disease secondary to cancer treatment. This will in turn improve quality of life and reduced morbidity and mortality.

Methods Subjects Postmenopausal women age 50-75 years diagnosed with EBC stage I-III eligible to receive (neo-)adjuvant chemotherapy or other adjuvant antineoplastic treatments Exclusion criteria include prior malignancy, preexisting T2D or other metabolic disease. The women will be recruited via the Department of Oncology at Rigshospitalet, Denmark.

Examinations

A cohort of 120 EBC women (WP1) will be followed from time of diagnosis through treatment and five years follow-up during AI treatment. Examinations will be performed either every six months or once a year, alongside routine visits and include:

WP1 (n=120)

* Blood samples (safety biochemistry, buffy coat (DNA), calcium homeostasis, bone markers, glucose, insulin and lipid levels, adipokines and inflammation markers
* Anthropometry (height, weight, waist/hip ratio)
* Neuropathy test by RR-interval-variation-analysis and vibration test
* Spirometry
* Questionnaires: food frequency (FFQ), physical activity (IPAQ)
* DXA scanning of body composition (GE Electric) and bone mass (Hologic)
* Urine
* App "Bone@BC"

Bone mineral density (BMD)/trabecular bone score (TBS) BMD is measured at the lumbar spine (mean of L2-L4), femoral neck and total hip on both sides using DXA (Hologic DiscoveryTM QDR Series scanner). DXA accurately determines 2 dimensional BMD (g/cm2) and detects patients at a heightened risk for osteoporotic fracture (23). The (unitless) calculated TBS is a novel, readily available, non-invasive clinical technique based on DXA images of the LS that provides a surrogate measure of the 3 dimensional microarchitecture of the skeleton (24). A high correlation between the TBS and CT42addressed microarchitecture has been observed (25), and the TBS is less influenced by the presence of osteoarthritis than BMD (26).

The same laboratory technician will perform all analyses. According to the manufacturer, the CV (coefficient of variation) of the total BMD is approximately 1% (Europe H. Hologic Osteoporosis Assesment. Reference Manual. 2006; Document No. Man-00214Revision 006).

Bone@BC app A newly developed app "Bone@BC" from RegionH that will be used by all women, is a guide and data collection app addressed to women with breast cancer receiving adjuvant anti-estrogen treatment. The app collects data on patient experiences (1. quality of life measures i.e. mobility, power/energy, mood, social contact and 2. measures of possible side-effects i.e. pain, dizziness, sleep) and from i.e. DXA-scanning, blood markers of bone turn-over and other biochemical measures. The specific data collection is for patient use, and can if approved by the patient, be part of the patient-caretaker-MD collaboration within the confines of this research study. The Bone@BC app will, with regard to patients in the study, only collect data for use in the study. The Bone@BC app has approved integration of app data with Region Security Requirements and is an official RegionH App legally approved at all levels (Nem-ID login, informed consent, approved by Datatilsynet).

Biological material Blood samples: Blood samples are obtained via venipuncture and processed at the central laboratory following routine procedures at Rigshospitalet.

Five ml urine will be stored in the biobank for metabolomics analysis.

Research biobank The biological material will be used for molecular analyses as described in the present protocol. These analyses including statistics will take place in a 10-year period after initiation of the project. After 10 years the biological material will be transferred to a research biobank at Rigshospitalet for future metabolic research. Participants will be made aware of this in the information material. The use of these samples would require re-approval of the Research Ethics Committee of the Capital Region. The establishment of a biobank has been approved by the Data Protection Agency.

Statistical considerations Based on literature studies the large cohort is estimated to include 120 enrolled EBC patients based on a power calculation of 80 finalizing the study (drop-out rate ~33% at year 5).

Side effects, risks and inconveniences During the examinations, there will be a temporary discomfort when applying peripheral venous catheters (venflon). In addition, blood tests are always associated with a risk of infection. All tissue samples will be excised by a trained professional, and the research team has comprehensive experience with blood and tissue sampling.

The total blood loss at each examination will not exceed 20 ml. Radiation from the DXA scan (DXA, TBS and Vertebral Fracture Assessment) is equivalent to 0.06 mRem and considered quite harmless. In comparison, a conventional X-ray image of the heart and lungs has a beam volume of approx. 30 mRem (0.3 mSv), and the annual background radiation in Denmark is about 300 mRem (3 mSv), corresponding to 0.8 mRem (0.008 mSv) daily.

If for any unforeseen reason, doubt arises about the health and security of the subject the study will be terminated immediately.

G. Data security All personal information regarding the participants will be protected by the "Lov om behandling af personlige oplysninger og Sundhedsloven". The protocol will be performed in accordance with the Declaration of Helsinki II, and has been approved by the Data Protection Agency. Analysis of biological material can possibly take place in Europe and/or in the United States. In such cases, the analyses will be conducted under the receiving country's laws and regulations, and in accordance with "Lov om behandling af personoplysninger".

Patient files will be used to check standard biochemistry tests. In addition due to the long observation period and the potential for relapse due to the underlying condition, it will be necessary to check patient files to maintain the security of the patients. Therefore consent from the patient will give the involved researchers access to the electronic patient files.

H. Financing Senior scientist, PhD. Charlotte Brøns and professor, dr.med. Peter Schwarz are responsible for initiating the research project. Neither have any conflicts of interest to declare.

Compensation There will not be given any compensation to patients participating in the study.

Recruitment All subjects will be recruited consecutively from the Department of Oncology, the breast cancer section, at Rigshospitalet, Denmark until 120 EBC patients have been included. All information given before consent is signed, will be to a researcher.

Publication and dissemination strategy The scientific results obtained from the study, whether positive, negative or inconclusive, will be written up in original manuscripts to become submitted to peer-reviewed international journals in the field. The results will furthermore be disseminated in oral presentations as well as in poster forms at relevant national and international meetings.

Ethical considerations Before entering the study, all individuals will receive oral and written information, and there will be a written consent to participate in the study. A unique subject ID number will be subscribed to all participants to anonymize data. The identification key (ID to personal information) will be encrypted and stored securely and separately from the unique ID number on a secure database, to ensure that no information on the participant can be assigned to the ID number. All data will automatically be backed up on a secure server. Only the research team will have access to the data. Neither the absolute nor the relative risk will be of unjustifiable size or of irresponsible character considering the impact of the study. The participants will gain information about personal health status. The current study provides an innovative and highly promising study approach to understanding metabolic and bone changes after adjuvant cancer treatments in early non-metastatic breast cancer.

If necessary, participants are covered by the insurance of Rigshospitalet.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* Breast cancer stage I-III
* Eligible to receive (neo-)adjuvant chemotherapy/other antineoplastic treatment

Exclusion Criteria:

* Prior malignancy
* Metabolic disease (diabetes mellitus etc)

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women age 50-70 years diagnosed with breast cancer stage I-III eligible to receive (neo-)adjuvant chemotherapy or other adjuvant antineoplastic treatments including trastuzumab and CKK4-6 inhibitors, AI and bisphosphonate. Exclusion criteria include prior malignancy, preexisting T2D or other metabolic disease. The women will be recruited via the Department of Oncology at Rigshospitalet, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Bone Mineral Density | 1-5 years
  Change in bone mineral density
Metabolic syndrome | 1-5 years
  Change in number of patients with the metabolic syndrome

SECONDARY OUTCOMES:
Bone fracture | 1-5 years
  Change in number of fractures
Insulin resistance | 1-5 years
  Change in insulin resistance
Glucose | 1-5 years
  Change in blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schwarz, Prof, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nissen MJ, Shapiro A, Swenson KK. Changes in weight and body composition in women receiving chemotherapy for breast cancer. Clin Breast Cancer. 2011 Mar;11(1):52-60. doi: 10.3816/CBC.2011.n.009. PMID 21421523
- [Background] Dieli-Conwright CM, Wong L, Waliany S, Bernstein L, Salehian B, Mortimer JE. An observational study to examine changes in metabolic syndrome components in patients with breast cancer receiving neoadjuvant or adjuvant chemotherapy. Cancer. 2016 Sep 1;122(17):2646-53. doi: 10.1002/cncr.30104. Epub 2016 May 24. PMID 27219902
- [Background] Demark-Wahnefried W, Winer EP, Rimer BK. Why women gain weight with adjuvant chemotherapy for breast cancer. J Clin Oncol. 1993 Jul;11(7):1418-29. doi: 10.1200/JCO.1993.11.7.1418. PMID 8315439
- [Background] Guinan EM, Connolly EM, Healy LA, Carroll PA, Kennedy MJ, Hussey J. The development of the metabolic syndrome and insulin resistance after adjuvant treatment for breast cancer. Cancer Nurs. 2014 Sep-Oct;37(5):355-62. doi: 10.1097/NCC.0b013e3182a40e6d. PMID 24088604
- [Background] Peairs KS, Wolff AC, Olsen SJ, Bantug ET, Shockney L, Kantsiper ME, Carrino-Tamasi E, Snyder CF. Coordination of care in breast cancer survivors: an overview. J Support Oncol. 2011 Nov-Dec;9(6):210-5. doi: 10.1016/j.suponc.2011.06.008. PMID 22055890
- [Background] Ewertz M, Jensen MB, Gunnarsdottir KA, Hojris I, Jakobsen EH, Nielsen D, Stenbygaard LE, Tange UB, Cold S. Effect of obesity on prognosis after early-stage breast cancer. J Clin Oncol. 2011 Jan 1;29(1):25-31. doi: 10.1200/JCO.2010.29.7614. Epub 2010 Nov 29. PMID 21115856
- [Background] Goodwin PJ, Ennis M, Bahl M, Fantus IG, Pritchard KI, Trudeau ME, Koo J, Hood N. High insulin levels in newly diagnosed breast cancer patients reflect underlying insulin resistance and are associated with components of the insulin resistance syndrome. Breast Cancer Res Treat. 2009 Apr;114(3):517-25. doi: 10.1007/s10549-008-0019-0. Epub 2008 Apr 25. PMID 18437560
- [Background] Coskun T, Kosova F, Ari Z, Sakarya A, Kaya Y. Effect of oncological treatment on serum adipocytokine levels in patients with stage II-III breast cancer. Mol Clin Oncol. 2016 May;4(5):893-897. doi: 10.3892/mco.2016.815. Epub 2016 Mar 10. PMID 27123303
- [Background] Gadea E, Thivat E, Planchat E, Morio B, Durando X. Importance of metabolic changes induced by chemotherapy on prognosis of early-stage breast cancer patients: a review of potential mechanisms. Obes Rev. 2012 Apr;13(4):368-80. doi: 10.1111/j.1467-789X.2011.00957.x. Epub 2011 Dec 1. PMID 22133030
- [Background] Reid DM, Doughty J, Eastell R, Heys SD, Howell A, McCloskey EV, Powles T, Selby P, Coleman RE. Guidance for the management of breast cancer treatment-induced bone loss: a consensus position statement from a UK Expert Group. Cancer Treat Rev. 2008;34 Suppl 1:S3-18. doi: 10.1016/j.ctrv.2008.03.007. Epub 2008 Jun 2. PMID 18515009
- [Background] Chien AJ, Goss PE. Aromatase inhibitors and bone health in women with breast cancer. J Clin Oncol. 2006 Nov 20;24(33):5305-12. doi: 10.1200/JCO.2006.07.5382. No abstract available. PMID 17114665
- [Background] Amir E, Seruga B, Niraula S, Carlsson L, Ocana A. Toxicity of adjuvant endocrine therapy in postmenopausal breast cancer patients: a systematic review and meta-analysis. J Natl Cancer Inst. 2011 Sep 7;103(17):1299-309. doi: 10.1093/jnci/djr242. Epub 2011 Jul 9. PMID 21743022
- [Background] Becker T, Lipscombe L, Narod S, Simmons C, Anderson GM, Rochon PA. Systematic review of bone health in older women treated with aromatase inhibitors for early-stage breast cancer. J Am Geriatr Soc. 2012 Sep;60(9):1761-7. doi: 10.1111/j.1532-5415.2012.04107.x. PMID 22985145
- [Background] Shapiro CL, Manola J, Leboff M. Ovarian failure after adjuvant chemotherapy is associated with rapid bone loss in women with early-stage breast cancer. J Clin Oncol. 2001 Jul 15;19(14):3306-11. doi: 10.1200/JCO.2001.19.14.3306. PMID 11454877
- [Background] Coleman RE, Banks LM, Girgis SI, Kilburn LS, Vrdoljak E, Fox J, Cawthorn SJ, Patel A, Snowdon CF, Hall E, Bliss JM, Coombes RC; Intergroup Exemestane Study group. Skeletal effects of exemestane on bone-mineral density, bone biomarkers, and fracture incidence in postmenopausal women with early breast cancer participating in the Intergroup Exemestane Study (IES): a randomised controlled study. Lancet Oncol. 2007 Feb;8(2):119-27. doi: 10.1016/S1470-2045(07)70003-7. PMID 17267326
- [Background] Brufsky AM et al, Cancer 118, 398, 2012
- [Background] Coleman R, de Boer R, Eidtmann H, Llombart A, Davidson N, Neven P, von Minckwitz G, Sleeboom HP, Forbes J, Barrios C, Frassoldati A, Campbell I, Paija O, Martin N, Modi A, Bundred N. Zoledronic acid (zoledronate) for postmenopausal women with early breast cancer receiving adjuvant letrozole (ZO-FAST study): final 60-month results. Ann Oncol. 2013 Feb;24(2):398-405. doi: 10.1093/annonc/mds277. Epub 2012 Oct 9. PMID 23047045
- [Background] Griggs JJ, Liu Y, Sorbero ME, Jagielski CH, Maly RC. Adjuvant chemotherapy dosing in low-income women: the impact of Hispanic ethnicity and patient self-efficacy. Breast Cancer Res Treat. 2014 Apr;144(3):665-72. doi: 10.1007/s10549-014-2869-y. Epub 2014 Mar 5. PMID 24596046
- [Background] Ellis GK, Bone HG, Chlebowski R, Paul D, Spadafora S, Smith J, Fan M, Jun S. Randomized trial of denosumab in patients receiving adjuvant aromatase inhibitors for nonmetastatic breast cancer. J Clin Oncol. 2008 Oct 20;26(30):4875-82. doi: 10.1200/JCO.2008.16.3832. Epub 2008 Aug 25. PMID 18725648
- [Background] Ellis GK, Bone HG, Chlebowski R, Paul D, Spadafora S, Fan M, Kim D. Effect of denosumab on bone mineral density in women receiving adjuvant aromatase inhibitors for non-metastatic breast cancer: subgroup analyses of a phase 3 study. Breast Cancer Res Treat. 2009 Nov;118(1):81-7. doi: 10.1007/s10549-009-0352-y. Epub 2009 Mar 24. PMID 19308727
- [Background] Winters-Stone KM, Dobek J, Nail L, Bennett JA, Leo MC, Naik A, Schwartz A. Strength training stops bone loss and builds muscle in postmenopausal breast cancer survivors: a randomized, controlled trial. Breast Cancer Res Treat. 2011 Jun;127(2):447-56. doi: 10.1007/s10549-011-1444-z. Epub 2011 Mar 19. PMID 21424279
- [Background] Saarto T, Sievanen H, Kellokumpu-Lehtinen P, Nikander R, Vehmanen L, Huovinen R, Kautiainen H, Jarvenpaa S, Penttinen HM, Utriainen M, Jaaskelainen AS, Elme A, Ruohola J, Palva T, Vertio H, Rautalahti M, Fogelholm M, Luoto R, Blomqvist C. Effect of supervised and home exercise training on bone mineral density among breast cancer patients. A 12-month randomised controlled trial. Osteoporos Int. 2012 May;23(5):1601-12. doi: 10.1007/s00198-011-1761-4. Epub 2011 Sep 3. PMID 21892676
- [Background] Theodorou DJ, Theodorou SJ, Sartoris DJ. Dual-energy X-ray absorptiometry in diagnosis of osteoporosis: basic principles, indications, and scan interpretation. Compr Ther. 2002 Fall;28(3):190-200. doi: 10.1007/s12019-002-0028-6. PMID 12360631
- [Background] Silva BC, Bilezikian JP. Trabecular bone score: perspectives of an imaging technology coming of age. Arq Bras Endocrinol Metabol. 2014 Jul;58(5):493-503. doi: 10.1590/0004-2730000003456. PMID 25166040
- [Background] Dufour R, Winzenrieth R, Heraud A, Hans D, Mehsen N. Generation and validation of a normative, age-specific reference curve for lumbar spine trabecular bone score (TBS) in French women. Osteoporos Int. 2013 Nov;24(11):2837-46. doi: 10.1007/s00198-013-2384-8. Epub 2013 May 17. PMID 23681084
- [Derived] Marina D, Nielsen A, Buch-Larsen K, Andersson M, Rasmussen AK, Schwarz P. Impact of aromatase inhibitors on thyroid function in postmenopausal women with early-stage breast cancer: a prospective controlled study. Cancer Treat Res Commun. 2025;45:101020. doi: 10.1016/j.ctarc.2025.101020. Epub 2025 Oct 15. PMID 41172892
- [Derived] Lindholm A, Abrahamsen ML, Buch-Larsen K, Marina D, Andersson M, Helge JW, Schwarz P, Dela F, Gillberg L. Pro-inflammatory cytokines increase temporarily after adjuvant treatment for breast cancer in postmenopausal women: a longitudinal study. Breast Cancer Res. 2024 Oct 16;26(1):142. doi: 10.1186/s13058-024-01898-3. PMID 39415181
- [Derived] Christensen IB, Abrahamsen ML, Ribas L, Buch-Larsen K, Marina D, Andersson M, Larsen S, Schwarz P, Dela F, Gillberg L. Peripheral blood mononuclear cells exhibit increased mitochondrial respiration after adjuvant chemo- and radiotherapy for early breast cancer. Cancer Med. 2023 Aug;12(16):16985-16996. doi: 10.1002/cam4.6333. Epub 2023 Jul 13. PMID 37439084